CLINICAL TRIAL: NCT00001049
Title: A Phase I Evaluation of the Safety and Toxicity of Zidovudine and Didanosine in Combination in HIV-Infected or Exposed Infants and a Phase II Study of the Effect of Didanosine vs. Combination Therapy With Zidovudine and Didanosine on HIV-1 RNA in Infants With HIV Infection
Brief Title: A Study of Didanosine Use Alone or in Combination With Zidovudine in Infants Exposed to or Infected With HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 239; 11216 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To determine the pharmacokinetics, safety, and efficacy of didanosine (ddI) alone or in combination with zidovudine (AZT) in HIV-infected infants.

PER AMENDMENT 4/8/97: Part A study objectives are completed. Part B objectives: To assess the safety, toxicity, and tolerability and to compare anti-HIV activity, as measured by change in log10 RNA, of the two study arms.

Early treatment of HIV-infected infants with antiretroviral agents may prevent the early and rapid decline of CD4 count and immunologic function. Combination therapy may be preferred over monotherapy, since resistance to a single agent can develop rapidly. Currently, there is little information on ddI monotherapy in young infants less than 90 days and no information on the use of combination therapy in this population.

DETAILED DESCRIPTION:
Early treatment of HIV-infected infants with antiretroviral agents may prevent the early and rapid decline of CD4 count and immunologic function. Combination therapy may be preferred over monotherapy, since resistance to a single agent can develop rapidly. Currently, there is little information on ddI monotherapy in young infants less than 90 days and no information on the use of combination therapy in this population.

In Part A, a cohort of patients younger than 28 days (was less than 120 days; amended 6/20/95) of age receives open-label ddI monotherapy for 1 week before initiation of AZT/ddI combination therapy. After pharmacokinetic data are obtained, an additional cohort of patients receives ddI at a higher dose. An age-adjusted dose for ddI is determined for use in Part B. (NOTE: As of 2/13/95, Part A has completed accrued for infants 29 to 120 days of age.) Part B patients less than 90 days of age (was less than 180 days of age; amended 6/20/95) are randomized, on a double-blind basis, to receive ddI or AZT/ddI. All patients continue treatment until 12 months after the last patient on Part B is enrolled. PER AMENDMENT 4/8/97: Part A of this protocol is closed with accrual objectives met. Part B of the study will remain open for patient accrual until 6/2/97. Part B is designed as a 2-arm, randomized, double-blind study to assess safety, toxicity and tolerability as well as anti-HIV activity of ddI or AZT/ddI.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* PCP prophylaxis.

Allowed:

* Acetaminophen if not on a continual basis.

NOTE:

* Drugs that are metabolized by hepatic glucuronidation or that are associated with occurrence of pancreatitis are allowed but should be used with caution.

Patients must have at least one of the following:

* Documented HIV infection.
* Been born to an HIV-infected woman and receiving AZT.

PER AMENDMENT 4/8/97:

* Number 2 above no longer required with closure of Part A of study.
* Patients must have signed, informed consent of parent or legal guardian.

PER 6/20/95 AMENDMENT, patients in Part A must be less than 28 days of age and those in Part B must be less than 90 days of age.

PER 7/7/94 AMENDMENT, patients in Part A were less than 120 days of age and those in Part B were less than 180 days of age.

NOTE:

* All patients must have been more than 34 weeks gestation at birth.

Prior Medication:

Allowed:

* Prior vaccine therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Pancreatitis.
* Clinically unstable condition.
* Current participation on a vaccine trial or, for Part A, a perinatal trial if of indeterminate infection status.

Concurrent Medication:

Excluded:

* Vaccine therapy.

Patients with the following prior condition are excluded:

* Pancreatitis at any time since birth.

Prior Medication:

Excluded in Part B patients only:

* More than 90 days of prior antiretroviral or immunomodulator therapy, exclusive of therapy received in utero.

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180
Dates: Study Completion 1998-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A Kovacs, Study Chair; R Husson, Study Chair
Locations (47):
- United States (45):
  - Univ of Alabama at Birmingham Schl of Med / Pediatrics, Birmingham, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - San Francisco Gen Hosp, San Francisco, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Denver, Denver, Colorado
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Palm Beach County Health Dept, Riviera Beach, Florida
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
  - Med College of Virginia, Richmond, Virginia
- Puerto Rico (2):
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] McKinney RE Jr. Ongoing and future trials of antiretroviral therapy in the pediatric AIDS clinical trials group (PACTG). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:173